CLINICAL TRIAL: NCT06753175
Title: Underwater Galvanic Stimulation by 4-Cell Bath on Lymphedema Post Mastectomy.
Brief Title: Underwater Galvanic Stimulation by 4-Cell Bath on Lymphedema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of Physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005390
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema
Keywords: Mastectomy
MeSH Terms: conditions — Lymphedema | interventions — Baths; carbohydrate-deficient transferrin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (CDT + Underwater Galvanic Stimulation group (Experimental): This group includes 30 patients who will receive underwater galvanic stimulation by 4-cell bath with CDT for 2 months (3times/week) in addition to their medical treatment.
  Interventions: Device: underwater galvanic stimulation by 4-cell bath; Other: Complete Decongestive Therapy (CDT):
- Group B (CDT group): (Active Comparator): This group includes 30 patients who will receive only CDT for 2 months (3times/week) in addition to their medical treatment.

INTERVENTIONS:
Device: underwater galvanic stimulation by 4-cell bath — Underwater Galvanic Stimulation:
  * Equipment: 4-cell bath
  * Procedure: Patients will immerse their affected limbs in the 4-cell bath. Electrical stimulation will be applied at a frequency of 15 Hz and intensity of 20 mA for 20 minutes, 3 times per week (Han et al. 2020).
  Arms: Group A (CDT + Underwater Galvanic Stimulation group
Other: Complete Decongestive Therapy (CDT): — Complete Decongestive Therapy (CDT):
  * Manual Lymphatic Drainage (MLD): 60 minutes per session, 3 days per week.
  * Compression Therapy: Multilayer bandaging applied after MLD.
  * Exercise: Specific exercises performed with compression in place.
  * Skin Care: Routine skin and nail care to prevent infections (Curlett et al. 2020).
  Arms: Group A (CDT + Underwater Galvanic Stimulation group

SUMMARY:
Sixty female patients with lymphedema post mastectomy, aged 30-55 years, will be selected from Minia Oncology Institute. The participants will be randomly distributed into two equal groups:

1. Group A (CDT + Underwater Galvanic Stimulation group):

   This group includes 30 patients who will receive underwater galvanic stimulation by 4-cell bath with CDT for 2 months (3times/week) in addition to their medical treatment.
2. Group B (CDT group):

This group includes 30 patients who will receive only CDT for 2 months (3times/week) in addition to their medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* ▪ Female patients with lymphedema post mastectomy

  * Aged 30-55 years
  * No history of cardiac or renal disease
  * No contraindications to electrotherapy
  * All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* ▪ Cardiac diseases.

  * Patients with active cancer
  * Patients with pacemakers or other implantable devices
  * Patients with a history of seizures or epilepsy

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Measuring pain intensity: | 2 months
  The Visual Analogue Scale (VAS) will be employed. This 10cm line, marked from "no pain"(zero) to "worst pain (10) imaginable," will be used to represent the pain continuum. Patients will be guided on how to interact with the VAS scale, ensuring clarity and ease of use.
Measuring the volume of a patient's upper limb: | 2 months
  Essential tools such as a flexible tape measure, marker pen or pencil, and a recording sheet will be collected. Measurements will be taken at specific anatomical landmarks every 4 cm, including the wrist, the midpoint of the forearm, and where the upper arm meets the shoulder. The tape measure will be applied snugly around the limb without tightening, ensuring consistency in tension. Both the affected and non-affected limbs will be measured for comparison, with a more than 10% volume increase indicating potential edem. Circumference measurements will be recorded to the nearest 0.1 cm without indenting the skin.
  The frustum of a cone formula will be used to estimate each arm segment's volume, with repeated measures for ongoing assessment.
Improvement in quality of life: | 2 months
  Assessed using the Lymphedema Quality of Life Questionnaire (LYMQOL).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt